CLINICAL TRIAL: NCT06801886
Title: Effect of Silymarin Supplementation on Graft Function and Early Post-transplant Complications
Brief Title: Silymarin's Advantage on Graft Effectiveness
Acronym: SAGE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, ass.prof., MD, Ph.D., University Hospital, Martin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TNO_UNM
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Posttransplant Diabetes Mellitus; Acute Graft Rejection; Biopsy Proven Acute Rejection; Antibody Mediated Rejection of Kidney Transplant; Arterial Hypertension, Chronic Kidney Disease
Keywords: silymarin; biopsy proven acute rejection; dnDSA; PTDM; protocolar biopsy; kidney transplantation
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients suplemented with placebo
  Interventions: Other: Placebo Supplementation
- Silymarin (Experimental): Patients suplemented with silymarin
  Interventions: Drug: Silymarine supplementation

INTERVENTIONS:
Drug: Silymarine supplementation — 900 mg of silymarin supplementation daily during the early post-transplant period, (for 30 days) under standard treatment.
  Arms: Silymarin
Other: Placebo Supplementation — Placebo supplementation during the early post-transplant period (30 days) under standard treatment
  Arms: Placebo

SUMMARY:
The study examines the impact of silymarin supplementation during the early post-transplant period, administering 900 g daily for 30 days under standard treatment. Subsequently, the investigators investigate its impact on graft function, as measured by eGFR (CKD-EPI equation), UACR or UPCR, the development of dnDSA, rejection changes, and histological changes in the 3-month biopsy protocol. At the same time, investigators will investigate the effect of silymarin on metabolic complications-PTDM, DLP, disorders of calcium-phosphate metabolism, and arterial hypertension in the post-transplant period-in comparison with the placebo group. At the same time, investigators will investigate the safety and tolerance of silymarin.

ELIGIBILITY:
Inclusion Criteria:

* First or second kidney transplant recipient
* Deceased or living donor kidney transplant
* Patients receiving standard immunosuppression regimen:
* Tacrolimus or cyclosporine + Mycophenolate mofetil + Corticosteroids
* Body Mass Index (BMI) 18-35 kg/m²
* Willingness to provide informed consent
* Ability to understand and comply with study procedures
* Stable medical condition without significant comorbidities

Exclusion Criteria:

* Multi-organ transplant recipients
* Recipients of ABO-incompatible or highly sensitized transplants
* Active infectious complications at the time of transplantation: HIV, Active hepatitis B or C, Active cytomegalovirus (CMV) infection
* Patients with known liver disease: Cirrhosis, Active hepatitis, ALT or AST > 2.5 times the upper limit of normal
* Significant cardiovascular disease: Recent myocardial infarction (within 6 months), Unstable angina, Severe heart failure (NYHA Class III or IV)
* Malignancy within the past 5 years (except successfully treated non-melanoma skin cancer)
* Current or recent (within 30 days) participation in another clinical trial
* Pregnancy or planned pregnancy during the study period
* Known allergy or hypersensitivity to silymarin or milk thistle
* Patients taking medications with significant interactions with silymarin:

Anticoagulants, Cytochrome P450 enzyme modulators

* Psychiatric conditions that may interfere with study compliance
* Uncontrolled diabetes mellitus (HbA1c > 8.5%)
* History of non-compliance with medical treatment
* Patients with known genetic disorders affecting drug metabolism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
eGFR improvement | 3 months
  Investigators estimate 1 month of silymarin supplementation may improve eGFR by 5 ml/min/1.73 m2 compared to palcebo at 3 months. Assuming a standard deviation of 10 ml/min/1.73 m2, a two-sided aplha of 0.005, and 80 % power, a sample size 64 participants per group is required.
Inicidence of biopsy proven acute rejection | 6 months
  Investigators assume - by supplementing silymarine the incidence of BPAR diagnosed by 3rd month protocolar biopsy, will be lower.

SECONDARY OUTCOMES:
Incidence of PTDM | 6 months
  Investigators asssume by supplementing silymarine, the incidence of PTDM diagnosed according to 2024 guidelines will be lower in observed period.
Incidence of dyslipidemia | 6 months
  Investigators asssume by supplementing silymarine, the incidence of hypercholesterolemia or dyslipidemia will be lower in observed period.
Improved graft function in participatns with delayed graft function | 6 months
  Investigators assume that in the group of patients with DGF, those supplemented with silymarine will have better eGFR and graft function during the observed period.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goli F, Karimi J, Khodadadi I, Tayebinia H, Kheiripour N, Hashemnia M, Rahimi R. Silymarin Attenuates ELMO-1 and KIM-1 Expression and Oxidative Stress in the Kidney of Rats with Type 2 Diabetes. Indian J Clin Biochem. 2019 Apr;34(2):172-179. doi: 10.1007/s12291-018-0735-0. Epub 2018 Feb 6. PMID 31092990
- [Background] Kaur G, Athar M, Alam MS. Dietary supplementation of silymarin protects against chemically induced nephrotoxicity, inflammation and renal tumor promotion response. Invest New Drugs. 2010 Oct;28(5):703-13. doi: 10.1007/s10637-009-9289-6. Epub 2009 Jul 10. PMID 19590824
- [Background] Mohammadi H, Hadi A, Arab A, Moradi S, Rouhani MH. Effects of silymarin supplementation on blood lipids: A systematic review and meta-analysis of clinical trials. Phytother Res. 2019 Apr;33(4):871-880. doi: 10.1002/ptr.6287. Epub 2019 Mar 5. PMID 30834633
- [Background] Voroneanu L, Nistor I, Dumea R, Apetrii M, Covic A. Silymarin in Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Diabetes Res. 2016;2016:5147468. doi: 10.1155/2016/5147468. Epub 2016 Jun 1. PMID 27340676